CLINICAL TRIAL: NCT03747393
Title: Exploring the Value of the Veterans Affairs (VA) and Department of Defense (DoD) Clinical Practice Guidelines for Non-Surgical Management of Knee Osteoarthritis in the Military Health System
Brief Title: Non-Surgical Management of Knee Osteoarthritis in the Military Health System (MHS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Dan Rhon, Director, Primary Care Musculoskeletal Research Center, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C2018.117d; W81XWH-18-1-0788 (Other Grant/Funding Number: DoD - Clinical Rehabilitation Medicine Research Program)
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; physical therapy; clinical practice guidelines; military service members; self-management
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness parallel-group randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DoD/VA CPG Core Set (Active Comparator): The standard core set of interventions recommended by the DoD/VA clinical practice guidelines for non-surgical management of knee OA.
  Interventions: Behavioral: DoD/VA CPG Core Set
- DoD/VA CPG Core Set + PT (Experimental): In addition to DoD/VA clinical practice guidelines, patients will be referred to physical therapy (PT). Physical therapy will consist of evidence-based interventions that can be provided by a PT (exercise, manual therapy, education).
  Interventions: Behavioral: DoD/VA CPG Core Set + PT; Behavioral: DoD/VA CPG Core Set

INTERVENTIONS:
Behavioral: DoD/VA CPG Core Set + PT — Participants randomized to receive the core set management class and physical therapy will be scheduled for their initial physical therapy evaluation approximately 1 week from their enrollment date. The purpose of the evaluation will be to identify relevant impairments that can be addressed during the physical therapy treatments. After this initial evaluation, the goal is for the patient to receive approximately 4 weeks of physical therapy (about 8-10 sessions in the clinic 2-3 times per week). Consistent with a pragmatic study we will not use placebos to blind patients or attempt to balance provider contact.
  Arms: DoD/VA CPG Core Set + PT
Behavioral: DoD/VA CPG Core Set — The published clinical practice guideline recommends early use of a core set of management strategies to include patient education about their condition and the role of obesity in disease progression, activity and lifestyle modification focusing on physical activity, and a therapeutic exercise program. Implementation of the core set is recommended prior to any referral for consultation about invasive procedures such as intra-articular injections or TKA surgery. All patients with knee pain will be scheduled to receive the core set management strategy class as a part of the usual care route.

SUMMARY:
This study will compare two different treatment approaches for the management of knee osteoarthritis (OA). All subjects will receive a standardized approach consistent with the core set of recommendation from the Department of Defense (DoD) and Veterans Administration (VA) Clinical Practice Guidelines for Non-Surgical Management of Knee Osteoarthritis. Follow-up will occur over a 1 year period.

DETAILED DESCRIPTION:
There are gaps between actual clinical practice and published guidelines for management of knee OA. The VA/DoD Clinical Practice Guidelines leaves open the question of the effectiveness and cost-effectiveness of early referral to PT alongside the core set of management strategies for patients with knee OA. Prior studies have failed to include robust cost-effectiveness analyses to understand the policy implications of a recommendation to routinely refer patients with knee OA to PT in addition to implementing the core set of recommended management strategies. A comparative effectiveness parallel-group randomized controlled clinical trial examining these questions will be extremely informative for future updates of the VA/DoD Practice Guideline.

The core components of the clinical practice guidelines include education on nutrition and the role of obesity in OA, as well as the role of physical activity and exercise. The physical therapy component will be based on best current evidence, and consist of manual therapy, education for self-management, and exercise.

ELIGIBILITY:
Inclusion Criteria:

* TRICARE eligible beneficiaries (active duty, dependents, and military retired) with a primary complaint of knee pain.
* Able to speak and read English well enough to provide informed consent, follow study instructions and independently answer the questionnaires/surveys.
* Able to attend treatment sessions for a 4-week period.
* Age 18-60 years old
* The subject had an initial care visit in the last 90 days with a chief complaint of knee pain, or is scheduled to have one within the week.
* Satisfies American College of Rheumatology (ACR) clinical criteria for diagnosis of knee OA for at least one knee.

Exclusion Criteria:

* In the last year, the subject has received any invasive interventions including injections (corticosteroid, hyaluronic acid, etc.) or surgery for their knee
* History of Total Knee Arthroplasty (TKA)
* Has previously received formal PT for the same knee (> 2 visits) in the last year
* Has consulted a surgeon for knee pain for either knee in the past year
* History of severe neurologic (e.g., stroke, Parkinson's disease, etc.) or other condition that prevents walking independently for at least 5 minutes or engaging in a physical activity/exercise program.
* Anyone leaving military service for other than regular retirement, pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury.
* Systemic disease that could otherwise be responsible for the subjects knee pain (e.g. rheumatoid arthritis, gout, or psoriatic arthritis), non-musculoskeletal conditions causing knee pain, personal history of neoplasm, current or recent knee joint infection, recent fall/trauma to knee, acute fracture of knee, lower extremity amputation, or other more likely primary musculoskeletal knee disorders (e.g. patellar tendinopathy, bursitis, runner's knee, etc.)
* Currently has a referral to orthopedics or physical therapy for a knee disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information Systems (PROMIS) - Physical Function | 2 years
  The PROMIS is managed and endorsed by the NIH, and will be based on the Computer Adaptive Test, which does not have a set number of questions but instead "adapts" the test and number of questions based on prior answers it receives.

SECONDARY OUTCOMES:
Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) | 2 years
  The WOMAC Osteoarthritis score, which consists of 24 questions, and 3 different subscales: pain (Q1-5), stiffness (Q6-7) and physical function (Q8-24)
Patient Acceptable Symptom Scale (PASS) | 2 years
  The PASS is a global, dichotomized single-item score indicating if patients are satisfied with the current state of their symptoms. This tool has been validated in patients with OA. The PASS asks the patient; "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" Response options are "yes" or "no".
EuroQoL (EQ-5D) | 2 years
  The EQ-5D is a generic quality of life questionnaire that will assess quality of life on a scale that can be referenced to other disease conditions. The EQ-5D covers 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has 3 response categories: level 1, "no problems"; level 2, "some problems"; and level 3, "inability or extreme problems." Responses are combined to give a 5-digit descriptive health state classification (e.g., 11222). The EQ-5D yields a total of 243 possible health states. Valuations for each health state are available. The EQ-5D is commonly used in economic evaluation of interventions and cost-effectiveness analysis.

OTHER OUTCOMES:
Healthcare Utilization from Electronic Medical Records (EMR) | 2 years
  Healthcare utilization will be extracted for all participants for the 2 year period following . enrollment. Drug prescriptions, medical procedures, and specialty referrals will be identified.
Credibility Expectancy Questionnaire (CEQ) | 2 years
  The CEQ, a 6-item self-report evaluating treatment credibility and expectations for improvement, will be assessed at baseline after treatment group assignment is revealed to provide descriptive information about participants' perceptions of their treatment assignment and optimism for improvement. The CEQ may be used as a covariate if perceptions differ meaningfully between groups as participants' initial perceptions of treatment credibility can impact outcomes.
Marcus 5 Item Exercise Self Efficacy Scale (MESE) | 2 years
  The MESE is a 5 item self report measure of exercise self efficacy with good validity and reliability. Higher scores reflect higher self efficacy. Participants rate their confidence in the ability to participate in regular exercise when faced with barriers and obstacles such as fatigue, vacation or poor weather.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Rhon, DSc, Principal Investigator — Brooke Army Medical Center
Locations (3):
- United States (3):
  - Brooke Army Medical Center, San Antonio, Texas
  - Wilford Hall Ambulatory Surgical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Data is proprietary to the US Defense Health Agency (DHA) and can be requested through a Data Sharing Agreement Application that must then be approved by the Data Privacy Board at DHA.

REFERENCES:
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] Uthman OA, van der Windt DA, Jordan JL, Dziedzic KS, Healey EL, Peat GM, Foster NE. Exercise for lower limb osteoarthritis: systematic review incorporating trial sequential analysis and network meta-analysis. BMJ. 2013 Sep 20;347:f5555. doi: 10.1136/bmj.f5555. PMID 24055922
- [Background] Abbott JH, Robertson MC, Chapple C, Pinto D, Wright AA, Leon de la Barra S, Baxter GD, Theis JC, Campbell AJ; MOA Trial team. Manual therapy, exercise therapy, or both, in addition to usual care, for osteoarthritis of the hip or knee: a randomized controlled trial. 1: clinical effectiveness. Osteoarthritis Cartilage. 2013 Apr;21(4):525-34. doi: 10.1016/j.joca.2012.12.014. Epub 2013 Jan 8. PMID 23313532
- [Background] Dhawan A, Mather RC 3rd, Karas V, Ellman MB, Young BB, Bach BR Jr, Cole BJ. An epidemiologic analysis of clinical practice guidelines for non-arthroplasty treatment of osteoarthritis of the knee. Arthroscopy. 2014 Jan;30(1):65-71. doi: 10.1016/j.arthro.2013.09.002. Epub 2013 Nov 28. PMID 24290788
- [Background] Deyle GD, Allison SC, Matekel RL, Ryder MG, Stang JM, Gohdes DD, Hutton JP, Henderson NE, Garber MB. Physical therapy treatment effectiveness for osteoarthritis of the knee: a randomized comparison of supervised clinical exercise and manual therapy procedures versus a home exercise program. Phys Ther. 2005 Dec;85(12):1301-17. PMID 16305269

DOCUMENTS (1):
  • Informed Consent Form (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT03747393/ICF_000.pdf